CLINICAL TRIAL: NCT00436553
Title: A 24-month Randomized, Double-masked, Controlled, Multicenter, Phase IIIB Study Assessing Safety and Efficacy of Verteporfin Photodynamic Therapy Administered in Conjunction With Ranibizumab Versus Ranibizumab Monotherapy in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Brief Title: Efficacy/Safety of Verteporfin Photodynamic Therapy and Ranibizumab Compared With Ranibizumab in Patients With Subfoveal Choroidal Neovascularization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBPD952A2308
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
Keywords: Age-related macular degeneration; AMD; choroidal neovascularization; verteporfin; ranibizumab
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Verteporfin; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Verteporfin With Standard Fluence Rate Plus Ranibizumab (Experimental): Patients received three consecutive monthly ranibizumab injections on Day 1 and at Months 1 and 2, and thereafter as needed at intervals of at least 30 days based on retreatment criteria. These patients also received verteporfin photodynamic therapy (PDT) with standard fluence (SF) rate on Day 1 and then as needed from Month 3 at intervals of at least 90 days based on the retreatment criteria. From month 3 onward, retreatments were determined based on study-specific retreatment criteria that included retinal thickness by Optical Coherence Tomography (OCT), sub-retinal hemorrhage evaluated by ophthalmoscopic examination, visual acuity assessed using Early treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and choroidal neovascularization (CNV) leakage assessed by fluorescein angiography (FA). Patients received sham intravitreal injections for the first 12 months if retreatment with ranibizumab was not warranted based on the retreatment criteria.
  Interventions: Drug: Verteporfin Photodynamic Therapy; Drug: Ranibizumab; Drug: Ranibizumab Placebo
- Ranibizumab Monotherapy (Active Comparator): Patients received monthly ranibizumab injections for 12 months and thereafter as needed based on the retreatment criteria. These patients were also administered verteporfin placebo infusion with sham PDT on Day 1 and then as needed from Month 3 at intervals of at least 90 days based on the retreatment criteria. Retreatments were determined based on study specific retreatment criteria that included retinal thickness by Optical Coherence Tomography (OCT), sub-retinal hemorrhage evaluated by ophthalmoscopic examination, visual acuity assessed using Early treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and choroidal neovascularization (CNV) leakage assessed by fluorescein angiography (FA).
  Interventions: Drug: Ranibizumab; Drug: Verteporfin Placebo
- Verteporfin With Reduced Fluence Rate Plus Ranibizumab (Experimental): Patients received three consecutive monthly ranibizumab injections on Day 1 and at Months 1 and 2, and thereafter as needed at intervals of at least 30 days based on retreatment criteria. These patients also received verteporfin PDT with reduced fluence (RF) rate on Day 1 and then as needed from Month 3 at intervals of at least 90 days based on the retreatment criteria. From month 3 onward, retreatments were determined based on study-specific retreatment criteria that included retinal thickness by Optical Coherence Tomography (OCT), sub-retinal hemorrhage evaluated by ophthalmoscopic examination, visual acuity assessed using Early treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and choroidal neovascularization (CNV) leakage assessed by fluorescein angiography (FA). Patients received sham intravitreal injections for the first 12 months if retreatment with ranibizumab was not warranted based on the retreatment criteria.
  Interventions: Drug: Verteporfin Photodynamic Therapy; Drug: Ranibizumab; Drug: Ranibizumab Placebo

INTERVENTIONS:
Drug: Verteporfin Photodynamic Therapy — After a 10-minute intravenous infusion of verteporfin at a dose of 6 mg/m^2 body surface area, verteporfin was activated by light application of 50 J/cm^2 (Standard Fluence rate) or 25 J/cm^2 (Reduced Fluence rate) to the study eye, begun 15 minutes after the start of the infusion.
  Other Names: Visudyne
  Arms: Verteporfin With Reduced Fluence Rate Plus Ranibizumab; Verteporfin With Standard Fluence Rate Plus Ranibizumab
Drug: Ranibizumab — Ranibizumab 0.5 mg administered as an intravitreal injection.
  Other Names: Lucentis
Drug: Verteporfin Placebo — To maintain masking, as a placebo for verteporfin photodynamic therapy, patients were administered a 10-minute intravenous infusion of 5% dextrose solution, followed by light application of 50 J/cm^2 to the study eye, begun 15 minutes after the start of infusion.
  Arms: Ranibizumab Monotherapy
Drug: Ranibizumab Placebo — To maintain masking, patients in the combination groups received sham intravitreal injections whenever retreatment with active Ranibizumab was not warranted based on the retreatment algorithm.
  Arms: Verteporfin With Reduced Fluence Rate Plus Ranibizumab; Verteporfin With Standard Fluence Rate Plus Ranibizumab

SUMMARY:
This study evaluated the effect of combination therapy with verteporfin photodynamic therapy and ranibizumab on visual acuity and anatomic outcomes compared to ranibizumab monotherapy and the durability of response observed in patients with choroidal neovascularization secondary to age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender age 50 years or older
* Subfoveal choroidal neovascularization (CNV) due to age-related macular degeneration (AMD)

Exclusion Criteria:

* Choroidal neovascularization due to causes other than AMD
* Prior treatment for neovascular AMD in the study eye

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2007-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (43):
- United States (36):
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Sacramento, California
  - West Coast Retina Medical Group Inc. - 185 Berry St. Suite 130, San Francisco, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, ‘Aiea, Hawaii
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Wichita, Kansas
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Paducah, Kentucky
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Grand Rapids, Michigan
  - Novartis Investigative SIte, Royal Oak, Michigan
  - Novartis Investigative Site, Williamsburg, Michigan
  - Novartis Investigative Site, Independence, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Toms River, New Jersey
  - Novartis Investigative Site, Lynbrook, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Beachwood, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, West Mifflin, Pennsylvania
  - Novartis Investigative Site, West Columbia, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Kingsport, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Fairfax, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Canada (7):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Ivey Eye Institute, Dr. Thomas Sheidow, London, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Montreal, Quebec

REFERENCES:
- [Derived] Kaiser PK, Boyer DS, Cruess AF, Slakter JS, Pilz S, Weisberger A; DENALI Study Group. Verteporfin plus ranibizumab for choroidal neovascularization in age-related macular degeneration: twelve-month results of the DENALI study. Ophthalmology. 2012 May;119(5):1001-10. doi: 10.1016/j.ophtha.2012.02.003. Epub 2012 Mar 22. PMID 22444829

RESULTS

PARTICIPANT FLOW:
Groups:
- Verteporfin SF + Ranibizumab: Patients received three consecutive monthly ranibizumab injections on Day 1 and at Months 1 and 2, and thereafter as needed at intervals of at least 30 days based on retreatment criteria. These patients also received verteporfin photodynamic therapy (PDT) with standard fluence (SF) rate on Day 1 and then as needed from Month 3 at intervals of at least 90 days based on the retreatment criteria. From month 3 onward, retreatments were determined based on study-specific retreatment criteria that included retinal thickness by Optical Coherence Tomography (OCT), sub-retinal hemorrhage evaluated by ophthalmoscopic examination, visual acuity assessed using Early treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and choroidal neovascularization (CNV) leakage assessed by fluorescein angiography (FA). Patients received sham intravitreal injections for the first 12 months if retreatment with ranibizumab was not warranted based on the retreatment criteria.
- Verteporfin RF + Ranibizumab: Patients received three consecutive monthly ranibizumab injections on Day 1 and at Months 1 and 2, and thereafter as needed at intervals of at least 30 days based on retreatment criteria. These patients also received verteporfin PDT with reduced fluence (RF) rate on Day 1 and then as needed from Month 3 at intervals of at least 90 days based on the retreatment criteria. From month 3 onward, retreatments were determined based on study-specific retreatment criteria that included retinal thickness by Optical Coherence Tomography (OCT), sub-retinal hemorrhage evaluated by ophthalmoscopic examination, visual acuity assessed using Early treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and choroidal neovascularization (CNV) leakage assessed by fluorescein angiography (FA). Patients received sham intravitreal injections for the first 12 months if retreatment with ranibizumab was not warranted based on the retreatment criteria.
Period: Overall Study
Arm/Group | Verteporfin SF + Ranibizumab | Verteporfin RF + Ranibizumab | Ranibizumab Monotherapy
Started | 104 (The table shows 12 month data. "Started" indicates Randomized set of population.) | 105 | 112
Completed | 91 (Completed the 12 month study phase.) | 93 | 102
Not Completed | 13 | 12 | 10
Not completed — Adverse Event | 4 | 3 | 4
Not completed — Death | 3 | 1 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verteporfin SF + Ranibizumab | Verteporfin RF + Ranibizumab | Ranibizumab Monotherapy | Total
Number analyzed (Participants) | 104 | 105 | 112 | 321
Age Continuous [Mean (Standard Deviation); unit: years] | 77.5 (8.42) | 77.4 (8.48) | 77.2 (7.97) | 77.3 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 53 | 75 | 192
  Male | 40 | 52 | 37 | 129

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best-corrected Visual Acuity (BCVA) of the Study Eye at Month 12
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increase in the VA score indicates improvement in visual acuity.
Time Frame: Baseline and Month 12
Population: The Full analysis set (FAS) consisting of all randomized patients that received at least one application of study drug and had at least one post-baseline assessment for BCVA in the study eye. Last observation carried forward (LOCF) was utilized.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Verteporfin SF + Ranibizumab | Verteporfin RF + Ranibizumab | Ranibizumab Monotherapy
Number analyzed (Participants) | 103 | 104 | 110
Letters
  Baseline | 53.7 (13.52) | 54.6 (12.78) | 54.8 (13.55)
  Month 12 | 59.0 (17.47) | 59.0 (18.03) | 63.0 (18.88)
  Change from baseline | 5.3 (15.66) | 4.4 (15.47) | 8.1 (15.09)

2. Secondary Outcome: Change From Baseline in Total Area of Leakage of the Study Eye at Month 12
Description: Total area of leakage of the study eye was assessed at the Central Reading Center (CRC) using Fluorescein angiography (FA).
Time Frame: Baseline and Month 12
Population: Full analysis set (FAS), observed data.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Verteporfin SF + Ranibizumab | Verteporfin RF + Ranibizumab | Ranibizumab Monotherapy
Number analyzed (Participants) | 67 | 66 | 78
mm^2
  Baseline | 6.654 (4.0956) | 6.211 (5.0618) | 6.931 (4.6473)
  Month 12 | 3.472 (4.2340) | 3.024 (4.0188) | 3.177 (4.9930)
  Change from Baseline | -3.182 (4.9729) | -3.187 (5.9744) | -3.753 (5.8005)

3. Secondary Outcome: Percentage of Patients With Fluorescein Leakage in the Study Eye at Month 12
Description: The percentage of patients with leakage of the study eye was assessed at the Central Reading Center (CRC) using Fluorescein angiography (FA).
Time Frame: Month 12
Population: Full analysis set (FAS), observed data.
Measure: Number; unit: Percentage of participants
Arm/Group | Verteporfin SF + Ranibizumab | Verteporfin RF + Ranibizumab | Ranibizumab Monotherapy
Number analyzed (Participants) | 67 | 66 | 79
Percentage of participants | 58.2 (0) | 54.5 (0) | 41.8 (0)

4. Secondary Outcome: Change From Baseline in Central Retinal Thickness at Month 12
Description: Optical coherence tomography was performed in the study eyes and the evaluations of the images were performed by the central reading center.
Time Frame: Baseline and Month 12
Population: Full analysis set (FAS), observed data.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Verteporfin SF + Ranibizumab | Verteporfin RF + Ranibizumab | Ranibizumab Monotherapy
Number analyzed (Participants) | 76 | 80 | 89
micrometer
  Baseline | 444.654 (137.7119) | 446.638 (129.5482) | 456.824 (153.4270)
  Month 12 | 292.921 (79.2733) | 305.719 (80.4508) | 284.586 (75.4892)
  Change from Baseline | -151.733 (135.6200) | -140.919 (128.0741) | -172.238 (166.6691)

5. Primary Outcome: Percent of Patients With a Treatment-free Interval of at Least 3 Months Following the Month 2 Visit
Description: The number of patients with a ranibizumab treatment-free interval, ie, no active ranibizumab treatments for at least 3 months duration (at least 2 consecutive monthly visits), anytime following the Month 2 ranibizumab treatment. Only active ranibizumab treatments were considered.
Time Frame: Month 2 up to Month 11
Population: Full analysis set (FAS) - Only the combination groups were analyzed. The percent of subjects with a ranibizumab treatment-free interval of at least 3 months duration following the Month 2 ranibizumab treatment was calculated using the subjects still in the study at Month 5.
Measure: Number; unit: Percent of participants
Arm/Group | Verteporfin SF + Ranibizumab | Verteporfin RF + Ranibizumab
Number analyzed (Participants) | 95 | 97
Percent of participants | 92.6 [85.4 to 97.0] | 83.5 [74.6 to 90.3]

ADVERSE EVENTS:
Time Frame: Cumulative up to Month 24
Description: The Safety set consisted of all patients who received at least one dose of study drug and had at least one post-baseline safety assessment. One patient was not treated as randomized. The safety data set includes patients as they were treated.
Arm/Group | Verteporfin SF + Ranibizumab | Verteporfin RF + Ranibizumab | Ranibizumab Monotherapy
Serious Adverse Events (participants affected / at risk) | 32/104 | 29/106 | 41/111
Other Adverse Events (participants affected / at risk) | 85/104 | 81/106 | 87/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Verteporfin SF + Ranibizumab (N=104) | Verteporfin RF + Ranibizumab (N=106) | Ranibizumab Monotherapy (N=111)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 3
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 2 | 6
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Choroidal infarction (Study eye) (Eye disorders) | 1 | 0 | 0
Eye pain (Study eye) (Eye disorders) | 0 | 0 | 1
Macular hole (Study eye) (Eye disorders) | 1 | 0 | 0
Macular oedema (Study eye) (Eye disorders) | 1 | 0 | 0
Retinal artery occlusion (Fellow eye) (Eye disorders) | 0 | 0 | 1
Retinal artery occlusion (Study eye) (Eye disorders) | 0 | 0 | 1
Retinal haemorrhage (Study eye) (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Study eye) (Eye disorders) | 4 | 1 | 3
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Iodine allergy (Immune system disorders) | 0 | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Endophthalmitis (Study eye) (Infections and infestations) | 1 | 0 | 2
Gangrene (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Labyrinthitis (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 4
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pacemaker complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colorectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 3
Alcoholism (Psychiatric disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Vascular insufficiency (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Verteporfin SF + Ranibizumab (N=104) | Verteporfin RF + Ranibizumab (N=106) | Ranibizumab Monotherapy (N=111)
Anaemia (Blood and lymphatic system disorders) | 1 | 7 | 5
Blepharitis (Study eye) (Eye disorders) | 6 | 3 | 5
Cataract (Fellow eye) (Eye disorders) | 4 | 4 | 6
Cataract (Study eye) (Eye disorders) | 6 | 6 | 8
Choroidal neovascularisation (Fellow eye) (Eye disorders) | 7 | 12 | 8
Conjunctival haemorrhage (Study eye) (Eye disorders) | 13 | 18 | 18
Eye pain (Study eye) (Eye disorders) | 22 | 14 | 14
Foreign body sensation in eyes (Study eye) (Eye disorders) | 6 | 2 | 5
Lacrimation increased (Study eye) (Eye disorders) | 6 | 6 | 10
Macular degeneration (Fellow eye) (Eye disorders) | 8 | 6 | 12
Macular oedema (Study eye) (Eye disorders) | 5 | 7 | 1
Maculopathy (Study eye) (Eye disorders) | 6 | 4 | 2
Myodesopsia (Study eye) (Eye disorders) | 2 | 11 | 10
Ocular hyperaemia (Study eye) (Eye disorders) | 8 | 4 | 8
Retinal haemorrhage (Fellow eye) (Eye disorders) | 6 | 5 | 7
Retinal haemorrhage (Study eye) (Eye disorders) | 7 | 9 | 8
Retinal oedema (Study eye) (Eye disorders) | 8 | 4 | 3
Visual acuity reduced (Fellow eye) (Eye disorders) | 5 | 6 | 2
Visual acuity reduced (Study eye) (Eye disorders) | 10 | 9 | 5
Vitreous detachment (Study eye) (Eye disorders) | 6 | 5 | 4
Constipation (Gastrointestinal disorders) | 3 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 6
Nausea (Gastrointestinal disorders) | 9 | 8 | 7
Fatigue (General disorders) | 0 | 3 | 7
Oedema peripheral (General disorders) | 4 | 3 | 6
Bronchitis (Infections and infestations) | 8 | 6 | 3
Nasopharyngitis (Infections and infestations) | 10 | 6 | 13
Sinusitis (Infections and infestations) | 5 | 8 | 6
Upper respiratory tract infection (Infections and infestations) | 11 | 10 | 7
Urinary tract infection (Infections and infestations) | 7 | 7 | 9
Corneal abrasion (Study eye) (Injury, poisoning and procedural complications) | 0 | 1 | 6
Fall (Injury, poisoning and procedural complications) | 7 | 4 | 9
Procedural pain (Study eye) (Injury, poisoning and procedural complications) | 1 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 7 | 5
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 1 | 1
Dizziness (Nervous system disorders) | 6 | 0 | 7
Headache (Nervous system disorders) | 7 | 5 | 7
Anxiety (Psychiatric disorders) | 2 | 5 | 7
Insomnia (Psychiatric disorders) | 3 | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 6 | 6
Hypertension (Vascular disorders) | 9 | 13 | 12
Hypotension (Vascular disorders) | 4 | 2 | 6

LIMITATIONS AND CAVEATS:
Shorten the study duration from 24 months to 12 months based on results of the European combination study MONT BLANC (CBPD952A2309).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or until the publication of the trial results in their entirety.